CLINICAL TRIAL: NCT04249960
Title: Sustain and Reinforce the Transition From Child to Adult Mental Health Care in Switzerland : A Monocentric Nested Cohort Randomized Controlled Trial: The SORT Study.
Acronym: SORT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Dr Marco Armando, Principal Investigator, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-0853
Record Dates: First submitted 2019-11-14; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Psychiatric Disorder; Transition
Keywords: adolescents; psychiatric disorders; CAMHS; AMHS; transition
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition as usual (No Intervention): Young people in this group will receive usual care and transition as usual, they will be our control group.
- Managed transition (Experimental): Young people in this group will do the managed transition, they will be our experimental group.
  Interventions: Behavioral: Managed transition

INTERVENTIONS:
Behavioral: Managed transition — Young people, their family and clinicians will receive transition guidelines and will be asked to follow them as much as possible.
  Arms: Managed transition

SUMMARY:
Disruption of care during transition from child and adolescent mental health (CAMHS) to adult mental health services (AMHS) may adversely affect the health and well-being of service users. Indeed, transition-related discontinuity of care is a major health and societal challenge today. Current evidences show that this transition is not always properly managed and that improving the transition process can have a positive impact on the health and wellbeing of young people. Nevertheless, data available are still inconsistent and only few studies investigated possible models aimed at improving and operationalize the transition. At present, no information concerning the transition in the Geneva Canton is available.

According to this lack of evidence, the current study aims at: 1) mapping the CAMHS/AMHS interface; 2) evaluating the longitudinal course and outcomes of adolescents approaching the transition boundary (TB) of their CAMHS; 3) determining the effectiveness of an experimental model of managed transition in improving outcomes, compared with usual care; 4) comparing these results with those of the EU funded MILESTONE study from several other European countries.

The investigators will recruit all patients aged ≥ 16 years and 6 months from the Geneva Canton in charge at CAMHS and they will follow them for up to 24 months. CAMHS will be instructed to provide all their service users at the time of transition either usual care or a novel service called "Managed Transition", which will include the use of a new decision support tool, the Transition Readiness and Appropriateness Measure (TRAM). A nested cohort Randomised Controlled Trial (ncRCT) design will be applied to divide patients into the two groups. The health and wellbeing of the young people will be assessed at baseline and then followed-up for 24 months to see whether they transition to AMHS or are discharged or referred to some other service. The investigators will then evaluate what impact the different transition experiences have on young people's health and wellbeing, and whether the process of Managed Transition has any benefits as compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* 1) provides valid written informed consent, or assent, if below the legal age of consent;
* 2) age is within 18 months of reaching the transition boundary of their CAMHS - during the trial recruitment period;
* 3) has a mental disorder defined by DSM-IV-TR, DSM-5 or ICD 10/11, or is under the regular care of CAMHS (if not yet diagnosed);
* 4) Has an IQ ≥ 70 as ascertained by previous standardized assessment or diagnosed by clinician, or no indication of intellectual impairment.

Exclusion Criteria:

* 1) does not provide valid written informed consent, or assent, if below the legal age of consent;
* 2) is younger than 18 months before the transition boundary of their CAMHS;
* 3) has intellectual impairment (IQ < 70) as ascertained by standardized assessment or diagnosed by clinician;
* 4) if not able to (or expected not to be able to) complete the questionnaires due to severe physical disabilities or language problems, even with assistance from family members or research assistant.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Patient's health status (need for care) | Before transition compared to after transition (18 months)
  Measured at each time point using the Health of the Nation Outcome Scale for Children and Adolescents (HoNOSCA) completed by a trained research assistant. Scores will be compared between first and last time point. HoNOSCA is 5 point scale going from 0 = not a problem, 1 = minor issue not requiring intervention, 2 = slightly problematic, 3 = moderately serious problem, 4 = serious to very serious problem, 9= unknown/not applicable. Scores are calculated by adding up all the subscales (9s are not counted) and a higher score means a worse outcome.

SECONDARY OUTCOMES:
Health of the Nation Outcome Scale for Children and Adolescents (HoNOSCA) self report | Baseline, 6, 12 and 18 months
  Self-report "need for care" status measured by the Health of the Nation Outcome Scale for Children and Adolescents
Transition Related Outcome Measure (TROM) | 6, 12 or 18 months
  Transition Related Outcome Measure to assess outcomes post-transition completed by the young person, parent/carer and clinician
Child Behavior Checklist (CBCL) or Adult Behavior Checklist (ABCL) | Baseline and 18 months
  Emotional and behavioral disturbances measured by the Achenbach System of Empirically Based Assessment (ASEBA) Child Behavior Checklist (CBCL) or Adult Behavior Checklist (ABCL) questionnaires (parent/carer version). CBCL targets young people until 17 and ABCL after 17.
Clinical Global Impression Scale (CGIS) | Baseline, 6, 12 and 18 months
  The Clinical Global Impression Scale completed by the clinician assesses patient's ilness severity
World Health Organisation's quality of life (WHOQOL-BREF) | Baseline and 18 months
  Young person's quality of life is measured by World Health Organisation's quality of life questionnaire. It is completed by the young person.
EuroQol generic quality of life questionnaire (5Q-5D-5L) | Baseline, 6, 12 and 18 months
  Quality Adjusted Life Years (QALYs) and cost effectiveness are assessed by EuroQol generic quality of life questionnaire completed by the young person.
On Your Own Feet - Transition Experience Scale (OYOF-TES) | 6, 12 or 18 months
  Transition experience and readiness assessed by On Your Own Feet - Transition Experience Scale completed by the young person and parent/carer only once at the time point right after transition
Barriers to Care (BtC) | 6, 12 and 18 months
  Barriers to care assessed by Barriers to Care checklist completed by the young person if he/she is not using the available services any more
Client Service Receipt Inventory (CSRI) | Baseline, 6, 12 and 18 months
  Service use assessed by a Client Service Receipt Inventory adapted from the Milestone study; completed by the young person
Health of the Nation Outcome Scale for Children and Adolescents (HoNOSCA) clinician version | Baseline, 6, 12, and 18 months
  Need for care and mental health status measured by Health of the Nation Outcome Scale for Children and Adolescents completed by a trained research assistant with information from the young person, parent/carer and clinician to ensure accuracy
Kiddie Schedule for Affective Disorders and Schizophrenia-Present State and Lifetime (K-SADS-PL) | Baseline and 18 months
  Kiddie Schedule for Affective Disorders and Schizophrenia-Present State and Lifetime Version for DSM-IV performed by a trained research assistant
Prodromal questionnaire (PQ-16) | Baseline and 18 months
  Prodromal questionnaire to assess prodromal symptoms filled by the young person as a self report
General Assessment Scale for Social Functioning (GASC) | Baseline and 18 months
  General Assessment Scale for Social Functioning assesses patients general functioning filled by the clinician
Reflective Functioning Questionnaire (RFQ and PRFQ) self-report and parent version | Baseline
  Reflective Functioning Questionnaire assesses mentalisation abilities filled by the young person and parent/carer (two versions)
Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) | Baseline
  Social abilities are measured by the Anticipatory and Consummatory Interpersonal Pleasure Scale self report and parent/carer version
Multidimensional Peer Victimization Scale-Revised (MPVS-R) | Baseline and 18 months
  Multidimensional Peer Victimization Scale-Revised assesses bullying as a self report
Coddington Life Event Scale (CLES) | Baseline, 6, 12 and 18 months
  Important life events is assessed by the Coddington Life Event Scale self-report
Perceived Stress Reactivity Scale (PSRS) | Baseline
  Young person's stress status is measured by the Perceived Stress Reactivity Scale self report

CONTACTS AND LOCATIONS:
Locations (1):
- University of Geneva, Geneva, Switzerland

REFERENCES:
- [Background] Waylen A, Wolke D. Sex 'n' drugs 'n' rock 'n' roll: the meaning and social consequences of pubertal timing. Eur J Endocrinol. 2004 Nov;151 Suppl 3:U151-9. doi: 10.1530/eje.0.151u151. PMID 15554900
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] McGorry PD. The specialist youth mental health model: strengthening the weakest link in the public mental health system. Med J Aust. 2007 Oct 1;187(S7):S53-6. doi: 10.5694/j.1326-5377.2007.tb01338.x. PMID 17908028
- [Background] McGorry P. Transition to adulthood: the critical period for pre-emptive, disease-modifying care for schizophrenia and related disorders. Schizophr Bull. 2011 May;37(3):524-30. doi: 10.1093/schbul/sbr027. PMID 21505119
- [Background] Pottick KJ, Bilder S, Vander Stoep A, Warner LA, Alvarez MF. US patterns of mental health service utilization for transition-age youth and young adults. J Behav Health Serv Res. 2008 Oct;35(4):373-89. doi: 10.1007/s11414-007-9080-4. Epub 2007 Nov 17. PMID 18026842
- [Background] Kataoka SH, Zhang L, Wells KB. Unmet need for mental health care among U.S. children: variation by ethnicity and insurance status. Am J Psychiatry. 2002 Sep;159(9):1548-55. doi: 10.1176/appi.ajp.159.9.1548. PMID 12202276
- [Background] Forbes A, While A, Ullman R, et al. A multi-method review to identify components of practice which may promote continuity in the transition from child to adult care for young people with chronic illness or disability. Report for the National Coordinating Centre for NHS Service Delivery and Organisation R & D (NCCSDO). London, UK: The Florence Nightingale School of Nursing and Midwifery, King's College, 2002.
- [Background] Kennedy A, Sloman F, Douglass JA, Sawyer SM. Young people with chronic illness: the approach to transition. Intern Med J. 2007 Aug;37(8):555-60. doi: 10.1111/j.1445-5994.2007.01440.x. PMID 17640188
- [Background] Kennedy P, Pugh R, Millar E. Towards managing the whole system of care and improving continuity of care. Psychiatric Bulletin, 29(7): 252-254, 2005
- [Background] Davis M. Addressing the needs of youth in transition to adulthood. Adm Policy Ment Health. 2003 Jul;30(6):495-509. doi: 10.1023/a:1025027117827. PMID 13677456
- [Background] Singh S P, Paul M, Islam Z, et al. Transition from CAMHS to adult mental health services (TRACK): a study of service organisation, policies, process and user and carer perspectives. 2010. Report for the national institute for health research service delivery and organisation programme (SDO Project 08/1613/117).
- [Background] Wilson A, Tuffrey A, McKenzie C, Street C. After the flood: young people's perspectives on transition. Lancet Psychiatry. 2015 May;2(5):376-378. doi: 10.1016/S2215-0366(15)00126-1. Epub 2015 Apr 28. No abstract available. PMID 26360268
- [Background] Paul M, Street C, Wheeler N, Singh SP. Transition to adult services for young people with mental health needs: A systematic review. Clin Child Psychol Psychiatry. 2015 Jul;20(3):436-57. doi: 10.1177/1359104514526603. Epub 2014 Apr 7. PMID 24711585
- [Background] Hovish K, Weaver T, Islam Z, Paul M, Singh SP. Transition experiences of mental health service users, parents, and professionals in the United Kingdom: a qualitative study. Psychiatr Rehabil J. 2012 Winter;35(3):251-7. doi: 10.2975/35.3.2012.251.257. PMID 22246124
- [Background] McDonagh JE, Viner RM. Lost in transition? Between paediatric and adult services. BMJ. 2006 Feb 25;332(7539):435-6. doi: 10.1136/bmj.332.7539.435. No abstract available. PMID 16497736
- [Background] Colver AF, Merrick H, Deverill M, Le Couteur A, Parr J, Pearce MS, Rapley T, Vale L, Watson R, McConachie H; Transition Collaborative Group. Study protocol: longitudinal study of the transition of young people with complex health needs from child to adult health services. BMC Public Health. 2013 Jul 23;13:675. doi: 10.1186/1471-2458-13-675. PMID 23875722
- [Background] Aebi M, Kuhn C, Metzke CW, Stringaris A, Goodman R, Steinhausen HC. The use of the development and well-being assessment (DAWBA) in clinical practice: a randomized trial. Eur Child Adolesc Psychiatry. 2012 Oct;21(10):559-67. doi: 10.1007/s00787-012-0293-6. Epub 2012 Jun 22. PMID 22722664
- [Background] Singh SP. Transition of care from child to adult mental health services: the great divide. Curr Opin Psychiatry. 2009 Jul;22(4):386-90. doi: 10.1097/YCO.0b013e32832c9221. PMID 19417667
- [Background] Suhrcke M, Pillas D, Selai C. Economic aspects of mental health in children and adolescents. Social Cohesion for Mental Wellbeing among adolescents: WHO, 43-64, 2008.
- [Background] Petrou S, Johnson S, Wolke D, Hollis C, Kochhar P, Marlow N. Economic costs and preference-based health-related quality of life outcomes associated with childhood psychiatric disorders. Br J Psychiatry. 2010 Nov;197(5):395-404. doi: 10.1192/bjp.bp.110.081307. PMID 21037217
- [Background] Copeland WE, Wolke D, Shanahan L, Costello EJ. Adult Functional Outcomes of Common Childhood Psychiatric Problems: A Prospective, Longitudinal Study. JAMA Psychiatry. 2015 Sep;72(9):892-9. doi: 10.1001/jamapsychiatry.2015.0730. PMID 26176785
- [Background] Relton C, Torgerson D, O'Cathain A, Nicholl J. Rethinking pragmatic randomised controlled trials: introducing the "cohort multiple randomised controlled trial" design. BMJ. 2010 Mar 19;340:c1066. doi: 10.1136/bmj.c1066. No abstract available. PMID 20304934
- [Background] Hayes RJ, Moulton LH. Cluster randomised trials: Chapman & Hall/CRC; 2009.
- [Background] Gowers SG, Harrington RC, Whitton A, Lelliott P, Beevor A, Wing J, Jezzard R. Brief scale for measuring the outcomes of emotional and behavioural disorders in children. Health of the Nation Outcome Scales for children and Adolescents (HoNOSCA). Br J Psychiatry. 1999 May;174:413-6. doi: 10.1192/bjp.174.5.413. PMID 10616607
- [Background] Achenbach, T.M. and L.A. Rescorla, Manual for the ASEBA school-age forms and profiles. 2001, Burlington, VT: University of Vermont, Research Center for Children, Youth and Families.
- [Background] Achenbach, T.M. and L.A. Rescorla, Manual for the ASEBA adult forms and profiles. 2003, Burlington, VT: University of Vermont, Research Center for Children, Youth and Families.
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Loewy RL, Pearson R, Vinogradov S, Bearden CE, Cannon TD. Psychosis risk screening with the Prodromal Questionnaire--brief version (PQ-B). Schizophr Res. 2011 Jun;129(1):42-6. doi: 10.1016/j.schres.2011.03.029. Epub 2011 Apr 20. PMID 21511440
- [Background] Guy W, editor. ECDEU Assessment Manual for Psychopharmacology. Rockville, MD: U.S. Department of Health, Education, and Welfare; 1976.
- [Background] Cornblatt BA, Auther AM, Niendam T, Smith CW, Zinberg J, Bearden CE, Cannon TD. Preliminary findings for two new measures of social and role functioning in the prodromal phase of schizophrenia. Schizophr Bull. 2007 May;33(3):688-702. doi: 10.1093/schbul/sbm029. Epub 2007 Apr 17. PMID 17440198
- [Background] Skevington SM, Sartorius N, Amir M. Developing methods for assessing quality of life in different cultural settings. The history of the WHOQOL instruments. Soc Psychiatry Psychiatr Epidemiol. 2004 Jan;39(1):1-8. doi: 10.1007/s00127-004-0700-5. PMID 15022040
- [Background] Coddington RD. The significance of life events as etiologic factors in the diseases of children. II. A study of a normal population. J Psychosom Res. 1972 Jun;16(3):205-13. doi: 10.1016/0022-3999(72)90045-1. No abstract available. PMID 5072914
- [Background] Fonagy P, Luyten P, Moulton-Perkins A, Lee YW, Warren F, Howard S, Ghinai R, Fearon P, Lowyck B. Development and Validation of a Self-Report Measure of Mentalizing: The Reflective Functioning Questionnaire. PLoS One. 2016 Jul 8;11(7):e0158678. doi: 10.1371/journal.pone.0158678. eCollection 2016. PMID 27392018
- [Background] Luyten P, Mayes LC, Nijssens L, Fonagy P. The parental reflective functioning questionnaire: Development and preliminary validation. PLoS One. 2017 May 4;12(5):e0176218. doi: 10.1371/journal.pone.0176218. eCollection 2017. PMID 28472162
- [Background] Gooding DC, Pflum MJ. The assessment of interpersonal pleasure: introduction of the Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) and preliminary findings. Psychiatry Res. 2014 Jan 30;215(1):237-43. doi: 10.1016/j.psychres.2013.10.012. Epub 2013 Oct 22. PMID 24210182
- [Background] Betts LR, Houston JE, Steer OL. Development of the Multidimensional Peer Victimization Scale-Revised (MPVS-R) and the Multidimensional Peer Bullying Scale (MPVS-RB). J Genet Psychol. 2015 Jan-Apr;176(1-2):93-109. doi: 10.1080/00221325.2015.1007915. Epub 2015 Mar 16. PMID 25775213
- [Background] Schlotz W, Yim IS, Zoccola PM, Jansen L, Schulz P. The Perceived Stress Reactivity Scale: measurement invariance, stability, and validity in three countries. Psychol Assess. 2011 Mar;23(1):80-94. doi: 10.1037/a0021148. PMID 21280954
- [Background] Nelson EC, Eftimovska E, Lind C, Hager A, Wasson JH, Lindblad S. Patient reported outcome measures in practice. BMJ. 2015 Feb 10;350:g7818. doi: 10.1136/bmj.g7818. No abstract available. PMID 25670183
- [Background] Chisholm D, Knapp MR, Knudsen HC, Amaddeo F, Gaite L, van Wijngaarden B. Client Socio-Demographic and Service Receipt Inventory--European Version: development of an instrument for international research. EPSILON Study 5. European Psychiatric Services: Inputs Linked to Outcome Domains and Needs. Br J Psychiatry Suppl. 2000;(39):s28-33. doi: 10.1192/bjp.177.39.s28. PMID 10945075
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Vanheusden K, Mulder CL, van der Ende J, van Lenthe FJ, Mackenbach JP, Verhulst FC. Young adults face major barriers to seeking help from mental health services. Patient Educ Couns. 2008 Oct;73(1):97-104. doi: 10.1016/j.pec.2008.05.006. Epub 2008 Jun 27. PMID 18584997
- [Background] van Staa A, Sattoe JN. Young adults' experiences and satisfaction with the transfer of care. J Adolesc Health. 2014 Dec;55(6):796-803. doi: 10.1016/j.jadohealth.2014.06.008. Epub 2014 Aug 19. PMID 25149686
- [Background] Preti A, Pisano A, Cascio MT, Galvan F, Monzani E, Meneghelli A, Cocchi A. Validation of the Health of the Nation Outcome Scales as a routine measure of outcome in early intervention programmes. Early Interv Psychiatry. 2012 Nov;6(4):423-31. doi: 10.1111/j.1751-7893.2011.00329.x. Epub 2012 Jan 8. PMID 22225572
- [Background] Tuomainen H, Schulze U, Warwick J, Paul M, Dieleman GC, Franic T, Madan J, Maras A, McNicholas F, Purper-Ouakil D, Santosh P, Signorini G, Street C, Tremmery S, Verhulst FC, Wolke D, Singh SP; MILESTONE consortium. Managing the link and strengthening transition from child to adult mental health Care in Europe (MILESTONE): background, rationale and methodology. BMC Psychiatry. 2018 Jun 4;18(1):167. doi: 10.1186/s12888-018-1758-z. PMID 29866202
- See also: UK Guidelines on transition in mental health — https://www.rcpsych.ac.uk/docs/default-source/improving-care/better-mh-policy/college-reports/college-report-cr182.pdf?sfvrsn=8662b58f_2
- See also: NICE Guidelines on transition in mental health — https://www.nice.org.uk/guidance/ng43/evidence/full-guideline-pdf-2360240173